CLINICAL TRIAL: NCT01489605
Title: Comparison of GlideScope Groove to Standard GlideScope for Orotracheal Intubation: A Non-inferiority Study
Brief Title: GlideScope Groove vs. Standard GlideScope: A Non-inferiority Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Device Withdrawn from market
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Timothy Turkstra, Staff Anesthesiologist and Associate Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18477
Record Dates: First submitted 2011-12-08; First posted 2011-12-09 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Intubation, Orotracheal
Keywords: Orotracheal intubation, videolaryngoscopy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GlideScope Groove (Experimental): Patients will be intubated using the GlideScope Groove device. (Verathon)
  Interventions: Device: GlideScope Groove
- Control: Standard GlideScope (Active Comparator): Control: Patients will be intubated using standard practice, a standard GlideScope (Verathon)
  Interventions: Device: Control: Standard GlideScope

INTERVENTIONS:
Device: GlideScope Groove — Patients will be intubated using the GlideScope Groove device. (Verathon)
  Other Names: Verathon
  Arms: GlideScope Groove
Device: Control: Standard GlideScope — Patients will be intubated using the standard GlideScope. (Verathon)
  Other Names: Varathon
  Arms: Control: Standard GlideScope

SUMMARY:
Patients presenting for elective surgery requiring orotracheal intubation will be randomized to being intubated with either the GlideScope Groove video-laryngoscope or the standard GlideScope video-laryngoscope.

DETAILED DESCRIPTION:
See above. The primary outcome is time to intubation.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient booked for elective surgery requiring orotracheal intubation.

Exclusion Criteria:

1. Any patient with cervical spine abnormalities.
2. Any patients with known or probable difficult airways.
3. Any patient requiring rapid sequence induction.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Duration of Intubation | Day 1
  Duration of Intubation - Mask removal to ETCO2 confirmation

SECONDARY OUTCOMES:
Ease of intubation | Day 1
  Ease of intubation as noted by operator (measured on a 100 mm Visual Analogue Scale)
Incidence of trauma | Day 1
  Incidence of trauma
Number of failures to intubate | Day 1
  Number of failures to intubate
Use of external laryngeal pressure | Day 1
  Use of external laryngeal pressure
Laryngoscopic grade distribution | Day 1
  Laryngoscopic grade distribution according to Cormack and Lehane classification
Sore Throat | Day 3
  Patients will be surveyed with respect to the incidence of post-operative sore throat.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Turkstra, MD, M. Eng, Principal Investigator — UWO
Locations (2):
- Canada (2):
  - London Health Sciences Center University Hospital, London, Ontario
  - London Health Sciences Centre Victoria Campus, London, Ontario